CLINICAL TRIAL: NCT03611660
Title: Does the Addition of Mindfulness Enhance BMI Outcomes in Obese Adolescents Enrolled in the Bright Bodies Weight Management Program?
Brief Title: Does Mindfulness Enhance BMI in Obese Adolescents Enrolled in the Bright Bodies Weight Management Program?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Friends of Yale New Haven Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000021532
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity, stress
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Lifestyle Program ONLY (Active Comparator): Participants will receive an evidence-based 12-week family-based pediatric obesity program.
  Interventions: Behavioral: Traditional Healthy Lifestyle Program
- Traditional Lifestyle Program PLUS Mindfulness (Experimental): Participants will receive an evidence-based 12-week family-based pediatric obesity program plus 6 sessions of mindfulness meditation instruction.
  Interventions: Behavioral: Traditional Healthy Lifestyle Program; Behavioral: Mindfulness Meditation Instruction

INTERVENTIONS:
Behavioral: Traditional Healthy Lifestyle Program — Twice weekly meetings that focus on nutrition and exercise for 12 weeks.
Behavioral: Mindfulness Meditation Instruction — Participants receive six mindfulness sessions.
  Arms: Traditional Lifestyle Program PLUS Mindfulness

SUMMARY:
Participants will be randomized to an evidence-based healthy lifestyle program alone or a healthy lifestyle program with mindfulness meditation added. The purpose of the study will be to determine if mindfulness improves BMI outcomes more than the program alone due to the stress-reduction benefits of mindfulness.

DETAILED DESCRIPTION:
The study will randomize 44 adolescents (aged 11-17 yo) with BMI >95th percentile to traditional Bright Bodies Healthy Lifestyle Program or Lifestyle Program plus mindfulness meditation (6 sessions within the 12-week program) (22 per group). The traditional program includes exercise two evenings per week and nutrition/behavior modification one evening per week for 12 weeks. Mindfulness session topics include breathing meditation, body scan meditation, mindful eating techniques, and identification of hunger verses satiation. The primary outcome measure with be (1) BMI, while secondary outcomes include changes in (2) percent body fat, (3) perceived stress scale (questionnaire), (4) physical stress (saliva cortisol levels), and (5) overall caloric intake (pre and post food records). After the 3 month intervention, participants will engage in post measures and be asked to return 6 months later (9 months) for longer-term follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI >95th percentile for gender & age
* English-speaking subject and parent/caregiver
* Parent/caregiver willing to participate in weight mgt program

Exclusion Criteria:

* BMI >40 <27
* Psychiatric disorder or medical condition that precludes participation in program
* Currently taking medication that causes weight gain or loss
* Involvement in co-existing weight management program
* A positive pregnancy test
* Plans on moving out of the Greater New Haven area within 9 months

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Change from baseline at 12 weeks
  Body Mass Index (BMI) will be calculated using the standard formula from participants' height and weight. BMI = (Weight in Pounds / (Height in inches x Height in inches)) x 703
Body Mass Index (BMI) | Change from baseline at 9 months
  Body Mass Index (BMI) will be calculated using the standard formula from participants' height and weight. BMI = (Weight in Pounds / (Height in inches x Height in inches)) x 703

SECONDARY OUTCOMES:
Percent Body Fat | Change from baseline at 12 weeks
  Tanita Body Fat Analyzer uses a foot-to-foot bioelectrical impedence to capture participant's percent body fat.
Percent Body Fat | Change from baseline at 9 months
  Tanita Body Fat Analyzer uses a foot-to-foot bioelectrical impedence to capture participant's percent body fat.
Perceived Stress Scale | Change from baseline at 12 weeks
  The Perceived Stress Scale is the most widely used psychological instrument for measuring the perception of stress. It is a 10-item likert questionnaire published by Mind Garden that asks about feelings and thoughts during the last month. PSS scores are obtained by reversing responses (i.e., 0=4) for positively stated items and leaving score as is for negatively stated items. An average score for this age group is 14.2, with higher scores indicating more stress. Our hypothesis is a greater change (lower scores at post) in the mindfulness group + traditional than traditional group alone.
Perceived Stress Scale | Change from baseline at 9 months
  The Perceived Stress Scale is the most widely used psychological instrument for measuring the perception of stress. It is a 10-item likert questionnaire published by Mind Garden that asks about feelings and thoughts during the last month. PSS scores are obtained by reversing responses (i.e., 0=4) for positively stated items and leaving score as is for negatively stated items. An average score for this age group is 14.2, with higher scores indicating more stress. Our hypothesis is a greater change (lower scores at post) in the mindfulness group + traditional than traditional group alone.
Physical Stress | Change from baseline at 12 weeks
  A physical indicator of stress is measured by saliva cortisol. We are using saliva swabs by Salimetrics. A normal range for saliva cortisol is 0.007-0.115 mcg/dL. Our hypothesis is a greater change (lowered) in the mindfulness + traditional group than the traditional group alone.
Physical Stress | Change from baseline at 9 months
  A physical indicator of stress is measured by saliva cortisol. We are using saliva swabs by Salimetrics. A normal range for saliva cortisol is 0.007-0.115 mcg/dL. Our hypothesis is a greater change (lowered) in the mindfulness + traditional group than the traditional group alone.
Caloric Intake | Change from baseline at 12 weeks
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.
Fat Intake | Change from baseline at 12 weeks
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.
Sugar Intake | Change from baseline at 12 weeks
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.
Caloric Intake | Change from baseline at 9 months
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.
Fat Intake | Change from baseline at 9 months
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.
Sugar Intake | Change from baseline at 9 months
  Calories, fat (grams), and added sugar (grams) will be measured by a 3-day food record entered into our Nutrition Data Software for Research (NDSR) Program. We will measure change and our hypothesis is that kcal, fat, and added sugar will be lower in the mindfulness + traditional group than the traditional group alone.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: weight management program website — http://brightbodies.org